CLINICAL TRIAL: NCT04876027
Title: Dulaglutide and Calorie Restrict Diet (CRD) in Overweight/Obese Patients With Polycystic Ovary Syndrome
Brief Title: GLP-1 RAs in Patients With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Principal Investigator, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLP-1RAs PCOS
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — dulaglutide; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLP-1 RAs and calorie restrict diet group (Experimental): Intervention with GLP-1 RAs and calorie restrict diet until reaching the target weight loss(7%)
  Interventions: Drug: GLP-1 RAs; Other: calorie restricted diet
- calorie restrict diet group (Active Comparator): Intervention with calorie restrict diet until reaching the target weight loss(7%)
  Interventions: Other: calorie restricted diet

INTERVENTIONS:
Drug: GLP-1 RAs — GLP-1 receptor agonist is a glucagon-like peptide 1 analog, which is related to improving blood sugar control, weight loss and appetite suppression, and reducing cardiovascular risk.
  Other Names: Dulaglutide
  Arms: GLP-1 RAs and calorie restrict diet group
Other: calorie restricted diet — Calorie restricted diet can improve insulin sensitivity, liver fat in patients with visceral obesity, and metabolism and hormone levels in obese women with PCOS.

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder, with a prevalence of 5% to 15% in premenopausal women. Patients with PCOS presents as abnormal menstruation, ovulation disorders and/or hyperandrogenemia, and often accompanied by insulin resistance and other metabolic abnormalities. Visceral fat dysfunction is an important factor in the onset of PCOS. GLP-1 receptor agonist is a glucagon-like peptide 1 analog, which is related to improving blood sugar control, weight loss and appetite suppression, and reducing cardiovascular risk. The purpose of this study was to compare whether the combined treatment of GLP-1 receptor agonists and calorie restrict diet reduced more visceral fat of overweight/obese patients with PCOS at the same weight loss (7%) compared with calorie restrict diet alone.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18- 45;
* Meet 2003 Rotterdam criteria;
* overweight/obesity,BMI≥24kg/m2.

Exclusion Criteria:

* any contraindication to dulaglutide (known or suspected hypersensitivity to dulaglutide or related products, previous acute pancreatitis or chronic pancreatitis, inflammatory bowel disease; personal history or family history of medullary thyroid carcinoma, or personal history of multiple endocrine neoplasia type 2)；
* treatment with any other drugs that may interfere with the trial, including traditional Chinese medicine, contraceptives, metformin, GLP-1RA or pioglitazone within the last 3 months；
* chronic kidney disease or severe liver dysfunction；
* malignant tumors；
* mental illness;
* pregnancy or lactation；
* inflammatory bowel disease;
* recent participation in other weight-loss research projects within the last 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
the change in visceral adipose tissue | until achievement of the weight loss target,an average of 12 weeks
  the change in visceral adipose tissue (pretreatment-post-treatment) after achievement of the weight loss target

SECONDARY OUTCOMES:
menstrual frequency | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  number of menstruation in a year
systolic blood pressure | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  systolic blood pressure (SBP), mmHg
diastolic blood pressure | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  diastolic blood pressure (DBP), mmHg
fasting plasma glucose | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  fasting plasma glucose (FPG), mmol/L
postprandial plasma glucose | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  postprandial plasma glucose (PPG), mmol/L
fasting insulin | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  fasting insulin (FINS), mU/L
postprandial insulin | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  postprandial insulin (PINS), mU/L
glycosylated hemoglobin A1c | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  glycosylated hemoglobin A1c (HbA1c), %
homeostasis model assessment of insulin resistance | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  homeostasis model assessment of insulin resistance (HOMA-IR)
alanine aminotransferase | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  alanine aminotransferase (ALT), U/L
aspartate aminotransferase | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  aspartate aminotransferase (AST), U/L
Total cholesterol | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  Total cholesterol (TC), mmol/L
Triglycerides | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  Triglycerides (TG), mmol/L
high-density lipoprotein cholesterol | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  high-density lipoprotein cholesterol (HDL-c), mmol/L
low-density lipoprotein cholesterol | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  low-density lipoprotein cholesterol (LDL-c), mmol/L
Creatinine | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  Creatinine (Cr), umol/L
serum uric acid | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  serum uric acid (SUA), umol/L
luteinizing hormone | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  luteinizing hormone (LH), IU/L
follicle-stimulating hormone | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  follicle-stimulating hormone (FSH), IU/L
pituitary prolactin | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  pituitary prolactin (PRL), mIU/L
total testosterone | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  total testosterone (TT), ng/ml
free testosterone | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  free testosterone (FT), pg/ml
Sex hormone binding globulin | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  Sex hormone binding globulin (SHBG), nmol/L
Androstenedione | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  Androstenedione (AD), ng/ml
dehydroepiandrosterone sulfate | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  dehydroepiandrosterone sulfate (DHEAS), ug/dl
controlled attenuation parameter | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  controlled attenuation parameter (CAP), dB/m
liver stiffness measurement | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  liver stiffness measurement (LSM), kPa
total body fat | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  percentage of total body fat, %
total body lean | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  percentage of total body lean, %
total fat mass | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  total fat mass, kg
total lean mass | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  total lean mass, kg
the change in subcutaneous adipose tissue | from randomization to the time of achievement of the weight loss target, an average of 12 weeks
  the change in subcutaneous adipose tissue (pretreatment-post-treatment) after achievement of the weight loss target

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr, Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People' Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No